CLINICAL TRIAL: NCT05382715
Title: Ulcerative Colitis in Subjects of Clinical Routine: A Four Year, Multicenter, Prospective, Non-Interventional Study to Evaluate Utilization, Effectiveness, and Quality of Life With Ozanimod
Brief Title: A Study to Evaluate the Utilization, Effectiveness, and Quality of Life of Ozanimod in Participants With Ulcerative Colitis
Acronym: COLIBRI
Status: Terminated | Type: Observational
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-027
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Colitis, Ulcerative
Keywords: Colitis, Ulcerative; Zeposia; Ozanimod; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — ozanimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Specified Dose on Specified Days
  Other Names: Zeposia®

SUMMARY:
The purpose of this study is to monitor the use, effectiveness and treatment persistence with Ozanimod (Zeposia®) as well as quality of life in participants undergoing treatment for moderate-to-severe ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Only Ozanimod (Zeposia®) naïve participants can be included into this prospective study
* Participants are suitable for therapy with Ozanimod (Zeposia®) according to the physician's recommendation (made before enrollment and independently of this Non-Interventional Study (NIS))
* Treatment with Ozanimod (Zeposia®) must be in-label and follow the approved Summary of Product Characteristics (SmPC)
* Participants must have confirmed diagnosis of moderate-to-severe Ulcerative Colitis

Exclusion Criteria:

* Participants that have previously been treated with Ozanimod (Zeposia®)
* Participants with mild Ulcerative Colitis (UC)
* Participants with a stoma
* Participants participating in other clinical trials
* Participants with a planned surgical intervention and hospitalization due to UC
* Participants with any contraindications specified in the current version of the SmPC

Other protocol-defined Inclusion/Exclusion Criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate-to-severe ulcerative colitis (UC) who initiate treatment with commercially available Ozanimod (Zeposia®) according to summary of product characteristics (SmPC) will be observed in a real-world setting in Germany over a 4-year period.
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Clinical Remission, defined by a partial Mayo Score (pMayo) of ≤1 plus an RBS=0 | At week 10

SECONDARY OUTCOMES:
Persistence of therapy during the study course measured by the number of participants who are on continuous treatment | Up to Week 52
Number of participants with Clinical Response | At Week 10 and Week 52
Number of participants with Clinical Remission | Up to Week 52
Number of participants with clinical remission at week 52 in patients who showed clinical response at week 10 | Up to Week 52
Treatment modalities measured by the Treatment Satisfaction Questionnaire for Medication - 9 items (TSQM-9) | Up to 1 Year
Patient's satisfaction with therapy measured by the TSQM-9 | Up to 1 Year
Time to discontinuation of treatment | Up to 1 Year
Change from baseline in Patient-Reported Outcomes (PROs) with regards to fatigue measured by the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Up to 1 Year
Change from baseline in PROs with regards to quality of life measured by the Short Inflammatory Bowel Disease Questionnaire (sIBDQ) | Up to 1 Year
Number of participants with Adverse Events (AEs) | Up to 1 Year
Number of participants with Corticosteroid (CS)-Free clinical response | Up to 1 Year
Number of participants with CS-Free clinical remission | Up to 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Berlin, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome